CLINICAL TRIAL: NCT07030296
Title: Effects of Sprint Training With and Without a Weighted Vest on Running Speed in Pre-adolescent Baseball Players
Brief Title: Effects of Sprint Training With and Without Weighted Vests on Speed in Youth Baseball Players
Acronym: SWIFT-BASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Principal Investigator, Édison Andrés Pérez Bedoya, PhD, Federal University of Vicosa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Tecnológico de Antioquia
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Youth Baseball Speed, Sprint Training, Weighted Vest, Change of Direction
Keywords: Sprint training, weighted vest, baseball, youth athletes, speed performance

STUDY DESIGN:
Intervention Model Description: This was a parallel-group randomized controlled trial. Participants (U-14 male baseball players) were randomly assigned to one of two groups: one group performed sprint training with a weighted vest (approximately 10% of body weight), and the other group performed the same sprint training protocol without a vest. The intervention included 16 training sessions over approximately 6 weeks. Sprint performance was measured before and after the intervention using 30-yard, 60-yard, and 60-yard change-of-direction tests. Randomization was conducted using simple random allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprint Training With Weighted Vest (Experimental): Participants in this arm performed sprint training while wearing a weighted vest equivalent to approximately 10% of their body weight. The program consisted of 16 sessions over six weeks and included linear sprints and change-of-direction drills. Sprint speed was assessed before and after the intervention.
  Interventions: Behavioral: Sprint Training With Weighted Vest
- Sprint Training Without Weighted Vest (Active Comparator): Participants in this group completed the same sprint training program as the experimental group but without wearing a weighted vest. The program lasted 16 sessions over approximately six weeks and included linear sprints and agility drills. Sprint performance was measured before and after the intervention.
  Interventions: Behavioral: Sprint Training Without Weighted Vest

INTERVENTIONS:
Behavioral: Sprint Training With Weighted Vest — Participants performed a sprint training program wearing a weighted vest equal to approximately 10% of their body weight. The program lasted 6 weeks and included 16 sessions of linear and change-of-direction sprint drills. The goal was to examine whether the added external load improved running speed over 30 and 60 yards.
  Other Names: Resisted Sprint Training
  Arms: Sprint Training With Weighted Vest
Behavioral: Sprint Training Without Weighted Vest — Participants completed the same sprint training program as the experimental group but without the use of a weighted vest. The intervention lasted 6 weeks and consisted of 16 sessions including sprint and agility exercises. This group served as the control condition to assess the effect of external resistance.
  Other Names: Unresisted Sprint Training
  Arms: Sprint Training Without Weighted Vest

SUMMARY:
Brief Summary We want to find out whether training with a weighted vest can help improve speed in U-14 baseball players. To do this, we will conduct a study with athletes like you, comparing performance before and after the training program.

How will we do it?

Participants will be randomly assigned to one of two groups:

Group 1: Will train with a weighted vest.

Group 2: Will train without a weighted vest.

Both groups will follow the same training program over 16 sessions. Running speed will be measured before and after the program to evaluate any improvements.

Who can participate?

Boys aged 13 to 14 years.

Members of the Tigres Baseball Club from San Pedro de Urabá.

Must have permission from a parent or legal guardian.

Who cannot participate?

Players with current injuries.

Those who regularly practice another sport.

Those who leave the club or are unable to complete the pre- and post-tests.

Is it safe? Yes! All procedures follow safety guidelines and will be conducted with informed consent from players and their families. Our goal is to enhance sports performance in a safe and effective way.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effects of sprint training with and without a weighted vest on running speed in male U-14 baseball players. The intervention will consist of a standardized sprint training program performed over 16 sessions (2-3 sessions per week for approximately 6 weeks). Participants will be randomly assigned into two groups: an experimental group using weighted vests and a control group without weighted vests.

The weighted vest will represent approximately 10% of the participant's body weight and will be worn during specific sprint training exercises. Both groups will perform the same sprint-based training protocol, including linear sprints and acceleration drills, under the supervision of qualified coaches.

The primary outcome will be sprint performance, assessed via time over 20 meters (with or without intermediate splits, depending on equipment availability). Measurements will be taken at baseline and after completion of the training program.

Inclusion and exclusion criteria have been defined to ensure participant safety and homogeneity of the sample. Ethical approval has been obtained, and informed consent will be secured from parents or legal guardians before participation. This study intends to contribute to evidence-based strategies for improving speed in youth baseball players through load-based sprint training interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged 13 to 14 years
* Member of the Tigres Baseball Club of San Pedro de Urabá
* Signed informed consent from parent or legal guardian
* Regular attendance at training sessions during the intervention period

Exclusion Criteria:

* Current musculoskeletal injury
* Regular participation in other sports or physical training programs
* Failure to complete pre- and post-intervention tests
* Withdrawal from the club during the study period

Ages: 13 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Change in 30-yard sprint time | Measured at baseline (pre-intervention) and after 16 training sessions (post-intervention), approximately 6 weeks apart.
  Time (in seconds) to complete a linear 30-yard sprint. Used to assess improvements in short-distance speed after the intervention.
Change in 60-yard sprint time | Pre- and post-intervention (6 weeks apart)
  Time (in seconds) to complete a 60-yard linear sprint. Assesses improvements in extended sprint speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Club de Baseball Tigers de San Pedro de Uraba, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request. De-identified data may be available to qualified researchers after publication of the main findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the main findings and will remain available for up to 3 years.
Access Criteria: De-identified individual participant data (IPD) will be available to qualified researchers upon reasonable request. Requests should include a brief research proposal and ethical approval (if applicable). Data will be shared via secure file transfer upon agreement with the principal investigator.